CLINICAL TRIAL: NCT00790387
Title: High Bolus Dose Tirofiban and Enoxaparin Provides Reduced Thrombin Generation and Inflammatory Markers in Patients With High Risk Undergoing Percutaneous Intervention
Brief Title: Tirofiban and Enoxaparin in High Risk Coronary Intervention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Prince Charles Hospital (Other Government)
Collaborators: Sanofi (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Assoc Professor Darren Walters, The Prince Chalres Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC2006
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2008-11

CONDITIONS: Acute Coronary Syndrome
Keywords: enoxaparin; tirofiban; percutaneous intervention; platelet inhibition; CD40L; Mac-1; prothrombin fragment 1+2.
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Enoxaparin; Tirofiban; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 High dose tirofiban and enoxaparin (Experimental): Enoxaparin was administered at the commencement of PCI at a dose of 0.75 mg/kg .
  Tirofiban was administered once the wire had crossed the lesion during PCI with a bolus dose of 25 µg/kg of bodyweight, followed by an infusion of 0.15 µg per kilogram per minute for 18 to 24 hours.
  Interventions: Drug: Enoxaparin
- 2 tirofiban and unfractionated heparin (Active Comparator): Tirofiban was administered once the wire had crossed the lesion during PCI with a bolus dose of 25 µg/kg of bodyweight, followed by an infusion of 0.15 µg per kilogram per minute for 18 to 24 hours.
  UFH heparin was administered as a bolus of 70 U/kg and additional heparin was given to maintain the activated clotting time (ACT) at 250
  Interventions: Drug: Tirofiban; Drug: unfractionated heparin

INTERVENTIONS:
Drug: Enoxaparin — Enoxaparin was administered at the commencement of PCI at a dose of 0.75 mg/kg
  Arms: 1 High dose tirofiban and enoxaparin
Drug: Tirofiban
  Arms: 2 tirofiban and unfractionated heparin
Drug: unfractionated heparin
  Arms: 2 tirofiban and unfractionated heparin

SUMMARY:
Patients undergoing coronary angioplasty are frequently treated with new drugs that stop blood platelets working and so improve the success of the procedure. Individual patients may vary in the dose of the drug required. New platelet tests have been developed which can be performed near the patient and possibly immediately tell the doctor the degree of platelet inhibition achieved so that the dose can be adjusted accordingly. This study aims to investigate if these platelet tests indicate if new anticoagulants are more effective at inhibiting platelet function than the traditional anticoagulants. The study will demonstrate if these newer drugs improve blood flow through the heart muscle and thereby provide better long term outcomes for patients undergoing percutaneous intervention.

DETAILED DESCRIPTION:
Objectives: The study assessed the benefit of high bolus dose tirofiban with enoxaparin compared to unfractionated heparin.

Introduction: The benefit of the use of glycoprotein IIb/IIa inhibitors with low molecular weight heparins in high risk patients undergoing percutaneous intervention (PCI) over traditional unfractionated heparin (UFH) is debated. Methods; The study is a prospective single center open-label trial of patients with high-risk acute coronary syndrome treated with PCI who were randomised to anticoagulation with UFH or enoxaparin with 'high dose' (25 mcg/kg bolus) tirofiban This study measured a panel of platelet activation markers, inflammatory biomarkers and thrombus generation between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients were recruited from those undergoing PCI with a planned placement of an intracoronary stent
* Including patients with unstable angina pectoris, acute coronary syndrome or NSTEMI
* Experienced ischaemic pain at rest
* Lasting 10 minutes and occurring within 7 days before enrollment
* As well as one of the following: ECG changes: New or presumably new ST-segment depression greater than or equal to 0.1 mV (1 mm), or transient (< 30 minutes) ST-segment elevation greater than or equal to 0.1 mV (1 mm) in at least 2 contiguous leads
* Abnormal cardiac enzymes within the 24 hours before enrollment, defined as elevated Troponin I defined as elevated Troponin I (above the normal reference -High-risk angiographic features that included intraluminal filling defect, angiographically visible thrombus eccentric lesion, type, location in a proximal major vessel and thrombolysis in myocardial infarction (TIMI) flow of II or less

Exclusion Criteria:

* Increased bleeding risk: ischaemic stroke within the last year or any previous haemorrhagic stroke, tumour or intracranial aneurysm;
* Recent (<1 month) trauma or major surgery (including bypass surgery);
* Active bleeding
* Unexplained clinically significant bleeding, thrombocytopenia (platelet count < 100 x 109/L) or history of thrombocytopenia with GP IIb/IIIa, heparin or enoxaparin therapy
* Angina from secondary causes such as severe uncontrolled hypertension (systolic blood pressure > 180 mm Hg despite treatment)
* Valvular disease, congenital heart disease, hypertrophic cardiomyopathy, -Thrombolytic therapy within preceding 24 hours
* Receiving antiIIb/IIIa therapy
* Creatinine clearance of <30 mL/min

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-06; Primary Completion 2005-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Thrombus generation as determined by Prothrombin fragment 1+2, D-dimer | 24 hours

SECONDARY OUTCOMES:
A panel of platelet activation markers:P selectin, MAC-1, PMAs, factor V/Va,Platelet inhibition as assessed by whole blood aggregometry | 10 minutes , 24 hours
Inflammatory biomarkers :CD40L,vWF and CRP | 10 minutes,24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Darren L Walters, Principal Investigator — The Prince Charles Hospital
Locations (1):
- The Prince Charles Hospital, Brisbane, Queensland, Australia